CLINICAL TRIAL: NCT04619628
Title: First-in-human, Randomised, Double-blind, Placebo-controlled, Dose-escalation Study in Healthy Young Adults Evaluating the Safety and Immunogenicity of COVI-VAC, a Live Attenuated Vaccine Candidate for Prevention of COVID-19
Brief Title: Safety and Immunogenicity of COVI-VAC, a Live Attenuated Vaccine Against COVID-19
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Codagenix, Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: CDX-CoV-001
Record Dates: First submitted 2020-11-05; First posted 2020-11-06 (Actual); Last update posted 2022-06-28 (Actual); Status verified 2022-06

CONDITIONS: COVID-19
Keywords: live attenuated; live attenuated vaccine; SARS-CoV-2; COVID-19
MeSH Terms: conditions — COVID-19 | interventions — COVI-VAC

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (7):
- Saline (Placebo Comparator): Normal saline
  Interventions: Other: Placebo
- Low dose cohort 1 (Experimental): COVI-VAC, single dose
  Interventions: Biological: COVI-VAC
- Medium dose cohort 1 (Experimental): COVI-VAC, single dose
  Interventions: Biological: COVI-VAC
- High dose cohort 1 (Experimental): COVI-VAC, single dose
  Interventions: Biological: COVI-VAC
- Low dose cohort 2 (Experimental): COVI-VAC, two doses 28 days apart
  Interventions: Biological: COVI-VAC
- Medium dose cohort 2 (Experimental): COVI-VAC, two doses 28 days apart
  Interventions: Biological: COVI-VAC
- High dose cohort 2 (Experimental): COVI-VAC, two doses 28 days apart
  Interventions: Biological: COVI-VAC

INTERVENTIONS:
Biological: COVI-VAC — intranasal, live attenuated vaccine against SARS-CoV-2
  Arms: High dose cohort 1; High dose cohort 2; Low dose cohort 1; Low dose cohort 2; Medium dose cohort 1; Medium dose cohort 2
Other: Placebo — normal saline
  Arms: Saline

SUMMARY:
This is the first study of COVI-VAC in humans. The purpose of the study is to evaluate the safety and immune response of COVI-VAC (a live attenuated vaccine to prevent COVID-19) in healthy adults aged 18 to 30 years. Approximately 48 participants will be enrolled into 1 of 3 dose groups (low, medium, high). Within each of these dose groups, participants will be assigned randomly to receive either 2 doses of COVI-VAC 28 days apart, 2 doses of placebo (saline), or 1 dose of COVI-VAC and 1 dose of placebo. COVI-VAC or placebo is administered by drops into each nostril. Neither the participants nor the researchers will know whether COVI-VAC or placebo has been received.

To assess the safety of the vaccine, each participant will record symptoms and oral temperature in a diary daily for 14 days after each dose. Safety laboratory tests, physical exams, ECGs, and a chest X-ray will also be performed, and peak expiratory flow and vital signs will be measured. Adverse events and medication use will be recorded.

Blood samples and intranasal samples will be collected to assess the immune response from the vaccine.

ELIGIBILITY:
Inclusion Criteria:

* Subjects who meet all of the following criteria may be included in the study:

  1. Men and women aged between 18 to 30 years of age, inclusive, on the day of signing the informed consent form (ICF)
  2. In good health with no history, or current evidence, of clinically significant medical conditions with particular reference to, but not restricted to, hypertension, diabetes, thromboembolic disorders, coronary heart disease, chronic obstructive lung disease, and no clinically significant test abnormalities that will interfere with subject safety, as defined by medical history, physical examination, vital signs (including oxygen saturation), ECG, spirometry, and safety laboratory tests as determined by the Investigator
  3. Total body weight of greater or equal to 50 kg and body mass index (BMI) greater or equal to 18.0 kg/m2 and less than or equal to 28.0 kg/m2 (the upper limit of the BMI may be increased to less than or equal to 30 kg/m2 at the Investigator's discretion in case of a muscular healthy subject for whom BMI may be biased upwards)
  4. Negative drugs of abuse, cotinine, and alcohol screen (unless explained by prescribed medication)
  5. Negative pregnancy test for women who have not been surgically sterilised
  6. Negative COVID Clear test

Exclusion Criteria:

Subjects who meet any of the following criteria will be excluded from the study:

1. Haemoglobin A1c ≥6.0% or 42 mmol/mol
2. Forced expiratory volume in 1 second (FEV1) less than 80% predicted value
3. Signs or symptoms suggestive of upper or lower respiratory tract infection (including fever or persistent cough) within 28 days of Day 1
4. Pregnant, possibly pregnant, or lactating women
5. Women who have been pregnant through the third trimester or given birth within the past 6 months
6. Planning a pregnancy (subject or partner) within 90 days after the last IMP dose
7. Inadequate venous access for repeated phlebotomy
8. History of confirmed or suspected SARS-CoV-2 infection
9. Contact with any individual subsequently confirmed to have SARS-CoV-2 within 14 days after contact
10. History of wheeze treated with inhaler(s)
11. Respiratory symptoms, including wheeze, that have ever resulted in hospitalisation
12. Known bronchial hyperreactivity to viruses
13. Any significant abnormality altering the anatomy of the nose in a substantial way or nasopharynx that may interfere with the aims of the study and in particular any of the nasal assessments or viral challenge (historical nasal polyps can be included, but large nasal polyps causing current and significant symptoms and/or requiring regular treatments in the last month are excluded)

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 48 (Actual)
Dates: Start 2020-12-11 (Actual); Primary Completion 2021-06-26 (Actual); Study Completion 2022-05-30 (Actual)

PRIMARY OUTCOMES:
Reactogenicity | 14 days after each dose
  Percentage of subjects with reactogenicity events
Adverse events | Days 1 through 57
  Percentage of subjects with adverse events
Serious adverse events | Days 1-400
  Percentage of subjects with serious adverse events

SECONDARY OUTCOMES:
IgG titre | Days 1, 15, 29, 43, 57, 120, 210, and 400
  IgG titre measured by ELISA in serum collected on Days 1, 15, 29, 43, 57, 120, 210, and 400
Neutralizing antibody titre | Days 1, 15, 29, 43, 57, 120, 210, and 400
  Neutralising antibody level measured by microneutralisation assay in serum

CONTACTS AND LOCATIONS:
Overall Officials: Daryl Bendel, MD, Principal Investigator — Hvivo
Locations (1):
- hVIVO, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No